CLINICAL TRIAL: NCT07036276
Title: Reducing and Breaking Up School-related Sedentary Behaviour Among Adolescents Using Co-creation
Acronym: G072223N
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Ghent (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ONZ-2025-0184
Record Dates: First submitted 2025-06-12; First posted 2025-06-25 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Sedentary Behaviour
Keywords: Adolescents; Youth; Student; School; Classroom; Sedentary behaviour; Participatory research; Co-creation; Co-adaptation

STUDY DESIGN:
Intervention Model Description: A three-arm clustered controlled trial will be conducted, including a co-adaptation intervention group, a standard intervention group and a control group. In September 2025, six schools will be recruited with immediate allocation to the 3 conditions. Pupils from Grade 7 and 8 will be informed about our study and provide an information letter for their parents. It will be specified that the co-adapted and standard intervention will be delivered to all adolescents as part of their curriculum, but that they are free to participate in the measurements. In September 2025 - January 2026, the co-adaptation process will take place in the co-adaptation intervention group. Between January and April 2026, the intervention will be implemented in the co-adaptation and standard intervention group. For the effect evaluation, there will be a pre-test after the co-adaptation process but before the implementation phase (January-February 2026), and a post-test after the implementation (March-April 2026).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Co-adaptation intervention group (Experimental): Co-adapted intervention: An existing co-created intervention will be adapted by researchers and 7th and 8th grade pupils and teachers during 3 to 5 design sessions in both co-adaptation intervention schools.
  Interventions: Behavioral: Co-adapted intervention
- Standard intervention group (Active Comparator): Standard intervention: The existing co-created intervention will be implemented in the standard intervention schools. So, adolescents and school staff from the standard intervention schools will not be involved in adapting the intervention.
  Interventions: Behavioral: Standard intervention
- Control group (No Intervention): No intervention will be implemented.

INTERVENTIONS:
Behavioral: Co-adapted intervention — An existing co-created intervention will be adapted by researchers and 7th and 8th grade pupils and teachers during 3 to 5 design sessions in both co-adaptation intervention schools.
  Arms: Co-adaptation intervention group
Behavioral: Standard intervention — The existing co-created intervention will be implemented in the standard intervention schools. So, adolescents and school staff from the standard intervention schools will not be involved in adapting the intervention.
  Arms: Standard intervention group

SUMMARY:
Adolescents spend the majority of the day sedentary, especially at school whilst sitting in class and at home when performing school-related tasks. As high levels of sedentary time are associated with adverse health effects, effective interventions are needed. To improve effectiveness, literature recommends a co-creative approach in which adolescents and other key stakeholders (such as teachers) are actively involved in the choice and development of intervention strategies. Therefore, this project aims to co-adapt a previously co-created intervention targeting adolescents' school-related sedentary behaviour. Further, the effect of this co-adapted intervention on adolescents' sedentary behaviour and related determinants, sleep, and mental wellbeing will be evaluated via a three-arm clustered controlled trial, including a co-adaptation intervention arm, a standard intervention arm (including schools that were not involved in co-adapting the intervention) and a control arm (continuing their curriculum as usual). By comparing these three arms, the investigators can evaluate the added value of co-creation compared to not involving adolescents or stakeholders in the development of an intervention. Lastly, the investigators will conduct a process evaluation of (1) the co-adaptation approach used to adapt the co-created intervention and (2) the implementation of both the co-adapted and standard interventions. Studies that evaluate co-created interventions are scarce. However, if such interventions prove to be more effective, this approach could be promising to change adolescents' health behaviour.

DETAILED DESCRIPTION:
1. Introduction This research project aims to co-adapt a co-created intervention targeting school-related sedentary behaviour. In this research, co-adaptation refers to the use of co-creation principles to adapt a co-created intervention to a new context (i.e., another school). The original intervention targeting school-related sedentary behaviour was co-created with Flemish secondary school pupils, teachers, and researchers in 2021-2022. In the current study, secondary school pupils and teachers from two schools, and researchers will be involved in the co-adaptation process. Next to co-adapting the intervention, this study aims to conduct an effect evaluation of the co-adapted intervention using a three-arm clustered controlled trial. Two schools will be allocated to each arm. In the first arm, the intervention will be co-adapted and implemented (co-adaptation intervention group); in the second arm, the original intervention will be implemented (standard intervention group); and the third arm is a control condition, which schools will continue their curriculum as usual. Finally, the investigators will conduct a process evaluation, which will evaluate (1) the co-adaptation process and (2) the implementation of the intervention in both the co-adaptation and standard intervention schools.
2. Participants Schools will be recruited in September 2025. The researcher will contact all secondary schools that are reachable within 40 minutes from the researcher's home town (Lier, Belgium) via e-mail and, if necessary, subsequently via telephone. If more than six schools show interest to participate, schools will be selected based on similar demographic characteristics (number of pupils and sex distribution) and education-related characteristics (such as the type of educational network). The focus of the study is on pupils and teachers in the first stage of secondary education (Grades 7 and 8, typically for ages 12-14). All pupils in these grades will be invited to participate in the study. A researcher will visit these classes to explain the study and distribute information and consent letters. Active consent will be asked from the pupils and at least one of their parents or legal representatives.
3. Procedure Between September 2025 and January 2026, the intervention will be co-adapted in the co-adaptation intervention schools. Researchers facilitating the co-adaptation process will complete a reflection form after each co-adaptation session with pupils and teachers to conduct a process evaluation of the co-adaptation process. In addition, focus groups with participating pupils and teachers will be conducted after the co-adaptation process. Before implementing the interventions in both intervention arms (co-adaptation intervention arm and standard intervention arm), a pre-test will be conducted in January-February 2026 in all six schools. From January to April 2026, the intervention will be implemented in both intervention arms over a six-week period. A post-test will be conducted after intervention implementation in March-April 2026. The pre-test and post-test will take place during school hours, at a time that is convenient for the school, in the presence of a researcher. During these visits, pupils will be given a GENEActiv to measure their sedentary and sleep time. They will then be asked to complete a questionnaire measuring determinants of reducing and regularly interrupting sedentary time and mental well-being. To evaluate intervention implementation, all pupils and teachers exposed to the intervention will be asked to complete an additional questionnaire during the post-test, supplemented by focus groups organised after the implementation. Further details on the measurements, are provided below.
4. Measurements

4.1. Process evaluation of the co-adaptation process and implementation of the interventions After each design session with pupils or teachers, researchers facilitating the session will complete a reflection form. These forms are used to reflect on the group process (e.g., if everyone participated) and the facilitators' role (e.g., if facilitators involved everyone). This way, facilitators can identify areas for improvement in subsequent sessions.

A trained female researcher with expertise in qualitative research will conduct 12 focus groups-6 with pupils and 6 with teachers. A second researcher will co-facilitate these focus groups and take notes. In the co-adaptation intervention schools, separate focus groups will be held with pupils and teachers after the co-adaptation process and after implementation. In the standard intervention schools, focus groups will be conducted only after the intervention has been implemented. At the start of each focus group, the interviewer will outline the goal of the focus group. Next, a semi-structured focus group will be conducted using an interview guide. Topics that will be discussed include: delivery (the extent to which the co-adaptation process and/or intervention was implemented as planned), participation (the level of engagement and participation of individuals or groups in the co-adaptation process and/or intervention), experience (subjective perceptions and evaluation of the co-adaptation process and/or intervention), context (social, cultural, economic, and political factors influencing the success or failure of the intervention), impact (the extent to which the co-adaptation process and/or intervention achieved its intended outcome(s), such as the impact on sedentary behaviour, but also the perceived impact on aspects such as pupils' classroom behaviour), and maintenance (the degree to which the relationships and/or outcomes formed during the co-adaptation process and/or intervention are sustained). Focus groups will be recorded and transcribed verbatim for analysis. In addition to the focus groups, a questionnaire will be administered to pupils and teachers after the implementation of the intervention, covering the delivery of the intervention and the participation of pupils in the intervention.

4.2 Effect evaluation Sedentary time and sleep duration will be measured using the GENEActiv accelerometer (ActivInsights Ltd., Kimbolton, UK), a waterproof tri-axial accelerometer (43 mm × 40 mm × 13 mm, 16 g). The accelerometer will be worn at the non-dominant wrist continuously over seven days using a 24-hour protocol. Data will be downloaded using the GENEActiv software and subsequently processed and analysed in R (R Development Core Team, 2010) using the GGIR package. Raw tri-axial acceleration values will be converted into a single omnidirectional measure of body acceleration using the Euclidean norm minus one (ENMO) metric. Data will then be reduced by averaging values over 1-second epochs. To determine physical activity intensity, the investigators will apply validated cut-points, classifying sedentary behaviour as values below 56.3 mg, light-intensity physical activity as values ranging from 56.3 to 191.6 mg, moderate-intensity physical activity as values between 191.6 and 695.8 mg, and vigorous-intensity physical activity as values exceeding 695.8 mg. Sedentary time and sedentary behaviour patterns, will be analysed across the entire day, during class hours, outside class hours (e.g., recess), and outside school hours.

To detect sleep, GGIR identifies periods of sustained inactivity. Sustained inactivity is defined as a period in which there is a change in arm angle of less than five degrees over a five-minute period. These thresholds have shown good accuracy for detecting sleep without the use of an activity diary compared to polysomnography, the gold standard sleep measure.

GGIR also estimates non-wear time by identifying periods of sustained low acceleration. Non-wear time will be determined when, for at least two out of three axes, the standard deviation of raw accelerometer data is less than 13 milligravity units (mg) and the data range is below 50 mg over 60-minute blocks, assessed every 15 minutes. GGIR provides two estimates to determine data validity: the number of valid hours and the fraction (%) of the night identified as invalid. In this study, the investigators will convert the fraction of the night identified as invalid to percentage of the night identified as valid (e.g., when 25% of the night is identified as invalid, this will be converted to 75% of the night identified as valid). Pupils will be included if they have at least 9 valid hours on four days for the sedentary time analysis, and at least 50% valid sleep data for five nights for the sleep duration analysis.

Next to the GENEActiv accelerometer, pupils will complete a questionnaire including items on determinants of reducing and regularly interrupting sedentary time in general (e.g., "I think it is important for my health to reduce my sitting time and to take regular breaks"), in the classroom (e.g., "I would rather sit in class than stand up"), and while making homework (e.g., "I prefer to do my schoolwork sitting down rather than standing up"). All items will be answered using a 5-point Likert scale (e.g., "totally disagree" to "totally agree"). Secondly, the questionnaire will assess adolescents' mental well-being using the World Health Organization-Five Well-Being Index (WHO-5). This scale consists of five statements relating to the past two weeks. Each statement is rated on a 6-point scale, with higher scores indicating better mental well-being.

ELIGIBILITY:
Inclusion Criteria:

* Secondary schools need to have at least 150 pupils in the first two grades (Grade 7 and 8).

Exclusion Criteria:

* None

Ages: 11 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 600 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Sitting time and patterns of sitting time | Assessed at baseline (pre-intervention) and immediately after the intervention period. The GENEActiv will be worn during one week.
  Sitting time and patterns of sitting time will be derived from a GENEActiv accelerometer that will be worn on the non-dominant wrist.
Determinants of reducing and regularly interrupting sedentary time in general, in the classroom, and while making homework | Assessed at baseline (pre-intervention) and immediately after the intervention period.
  These determinants will be measured using a questionnaire including items that will be answered on a 5-point Likert scale.

SECONDARY OUTCOMES:
Sleeping time | Assessed at baseline (pre-intervention) and immediately after the intervention period. The GENEActiv will be worn during one week.
  Sleeping time will be derived from a GENEActiv accelerometer that will be worn on the non-dominant wrist.
Mental well-being | Assessed at baseline (pre-intervention) and immediately after the intervention period.
  Mental well-being will be measured using the the World Health Organization-Five Well-Being Index (WHO-5).

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication.
Time Frame: The data will be published together with the publishing of manuscripts.
Access Criteria: This depends on the journal. The investigators will deposit the data into a data repository (i.e., OSF) or publish the data as supplementary file along with the manuscript in a journal.